CLINICAL TRIAL: NCT00732940
Title: A Phase 2, Multi-Center, Randomized, Open Label, Trial to Evaluate the Safety, Tolerability, and Biological Activity of 2 Dosing Schedules of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, Administered Subcutaneously to Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: Phase 2 Study of Belimumab Administered Subcutaneously to Subjects With Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated study for business reasons.
Sponsor: Human Genome Sciences Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGS1006-1070; 112232 (Other: GlaxoSmithKline)
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Systemic Lupus Erythematosus; Antibodies; Autoimmune Diseases; Belimumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belimumab Q2WKS (Experimental): Every other week: 100 mg of belimumab (1 injection) subcutaneous (under the skin) on days 0, 7, and 14, then every other week until final evaluation at Week 24 with option to continue receiving belimumab at the same dose through 144 week continuation period.
  Interventions: Drug: Belimumab 100 mg SC
- Belimumab 3X/WK (Experimental): Three times weekly: 200 mg of belimumab (2 injections of 100 mg each) subcutaneous (under the skin) on days 0, 2, and 4 then 100 mg three times a week until final evaluation at Week 24 with option to continue receiving belimumab at the same dose through 144 week continuation period.
  Interventions: Drug: Belimumab 100 mg SC

INTERVENTIONS:
Drug: Belimumab 100 mg SC — Belimumab 100 mg SC for 1 injection on Days 0, 7, 14, and then every two weeks.
  Other Names: LymphoStat-B™
  Arms: Belimumab Q2WKS
Drug: Belimumab 100 mg SC — Belimumab 100mg SC for 2 injections (of 100mg each) on Days 0, 2, and 4, then 100 mg (1 injection) three times per week.
  Arms: Belimumab 3X/WK

SUMMARY:
The purpose of this study is to test the safety and tolerability of repeated subcutaneous (SC) doses of belimumab in subjects with SLE.

DETAILED DESCRIPTION:
This clinical trial will evaluate the safety, pharmacokinetics (PK), and effect on biomarkers of repeated subcutaneous (SC) administration of belimumab in subjects with SLE. As data permit, an exploratory pharmacodynamic analysis will be performed to evaluate the correlation between belimumab serum exposure, PGA, SELENA SELDAI, and biomarker effects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria
* Active SLE disease
* On stable SLE treatment regimen

Exclusion Criteria:

* Pregnant or nursing
* Have received treatment with an B cell targeted therapy
* Have received treatment with a biologic investigational agent in the past year
* Have received intravenous (IV) cyclophosphamide within 180 days of Day 0
* Have severe lupus kidney disease
* Have active central nervous system (CNS) lupus
* Have required management of acute or chronic infections with the past 60 days
* Have current drug or alcohol abuse or dependence or within the past year
* Have a historically positive test or test positive at screening for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Have a history of an allergic or anaphylactic reaction to drugs, food, or insects requiring medical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Valerious Medical Group Research Center, Long Beach, California
  - Tampa Medical Group, PA, Tampa, Florida
  - Fiechtner Research, Inc., Lansing, Michigan
  - SUNY Downstate Medical Center, Brooklyn, New York
  - North Shore-LIJ Health System/Rheumatology, Allergy, Immunology, Lake Success, New York
  - Rheumatology Associates, Smithtown, New York
  - STAT Research, Inc., Dayton, Ohio
  - Oklahoma Center for Arthritis Therapy & Research, Tulsa, Oklahoma
  - Houston Institute for Clinical Research, Houston, Texas
- Hospital Central "Igancio Morones Prieto", San Lusi Potosi, Mexico

REFERENCES:
- [Derived] van Vollenhoven RF, Navarra SV, Levy RA, Thomas M, Heath A, Lustine T, Adamkovic A, Fettiplace J, Wang ML, Ji B, Roth D. Long-term safety and limited organ damage in patients with systemic lupus erythematosus treated with belimumab: a Phase III study extension. Rheumatology (Oxford). 2020 Feb 1;59(2):281-291. doi: 10.1093/rheumatology/kez279. PMID 31302695

RESULTS

PARTICIPANT FLOW:
Groups:
- Belimumab SC Q2WKS: 100 mg of belimumab (1 subcutaneous injection) on days 0, 7, and 14, then every other week until Week 24 with option to continue receiving belimumab at the same dose through 144 week continuation period.
- Belimumab SC 3X/WK: 200 mg of belimumab (2 subcutaneous injections of 100 mg each) on days 0, 2, and 4 then 100 mg three times a week until Week 24 with option to continue receiving belimumab at the same dose through 144 week continuation period.
Period: Overall Study
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Started | 28 | 28
Completed | 26 | 25
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK | Total
Number analyzed (Participants) | 28 | 28 | 56
Age Continuous [Mean (Standard Deviation); unit: years] | 39.2 (11.5) | 40.9 (13.1) | 40.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49
  Mexico | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Number of Participants Who Experienced Adverse Events (AEs) During the 24 Week Period.
Description: SEE ALSO ADVERSE EVENTS RESULTS SECTION
Time Frame: Up to 24 weeks
Population: Please see Adverse Events Section
Measure: Number; unit: Percentage of participants
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 28 | 28
Percentage of participants
  Percent of patients with at least 1 AE | 89.3 | 85.7
  Percent of patients with at least 1 Serious AE | 7.1 | 14.3
  Percent of patients with an AE resulting in death | 0 | 0

2. Secondary Outcome: Mean Serum Belimumab Concentration Levels (Pharmacokinetic [PK]) Over 24 Weeks.
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 28 | 26
µg/mL | 20.5 (11.6) | 120.8 (53.7)

3. Secondary Outcome: Absolute Change From Baseline in IgA at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 26 | 25
g/L | -0.3 (0.08) | -0.3 (0.10)

4. Secondary Outcome: Median Percent Change From Baseline in IgA at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 26 | 25
Percentage | -8.1 [-45.1 to 15.4] | -10.7 [-36.4 to 34.1]

5. Secondary Outcome: Absolute Change From Baseline in IgG at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
g/L | -2.2 (0.7) | -1.4 (0.7)

6. Secondary Outcome: Median Percent Change From Baseline in IgG at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
Percentage | -11.1 [-47.0 to 12.1] | -9.5 [-42.9 to 94.0]

7. Secondary Outcome: Absolute Change From Baseline in IgM at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: g/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
g/L | -0.3 (0.04) | -0.4 (0.07)

8. Secondary Outcome: Median Percent Change From Baseline in IgM at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
Percentage | -25.6 [-80.0 to 11.0] | -26.9 [-71.6 to 170.6]

9. Primary Outcome: Absolute Change From Baseline in CD20+ (Total) B Cells at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 23 | 23
cells/mm^3 | -53.5 (20.4) | -75.3 (23.6)

10. Primary Outcome: Median Percent Change From Baseline in CD20+ (Total) B Cells at Week 24.
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 23 | 23
Percentage | -33.5 (8.88) [-86.3 to 55.2] | -38.2 (13.26) [-86.3 to 130.8]

11. Primary Outcome: Absolute Change From Baseline in CD20+/CD27- (Naive) B Cells at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 23 | 23
cells/mm^3 | -81.9 (18.5) | -95.0 (20.8)

12. Primary Outcome: Median Percent Change From Baseline in CD20+/CD27-(Naive) B Cells at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 23 | 23
Percentage | -60.9 (6.47) [-89.6 to 4.8] | -66.7 (8.0) [-90.2 to 85.7]

13. Primary Outcome: Absolute Change From Baseline in CD20+/CD69+ (Activated) B Cells at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: cells/mL
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 24 | 23
cells/mL | 1100.3 (389.8) | -77.2 (456.9)

14. Primary Outcome: Median Percent Change From Baseline in CD20+/CD69+ (Activated) B Cells at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 24 | 23
Percentage | 45.2 [-69.6 to 1496.3] | 10.2 [-87.0 to 779.6]

15. Primary Outcome: Absolute Change From Baseline in CD20+/CD27+ (Memory) B Cells at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: cells/mm^3
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 23 | 23
cells/mm^3 | 27.7 (6.0) | 19.6 (6.2)

16. Primary Outcome: Median Percent Change From Baseline in CD20+/CD27+ (Memory) B Cells at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 23 | 23
Percentage | 84.2 [-37.5 to 288.9] | 100.0 [-45.5 to 600.0]

17. Secondary Outcome: Absolute Change From Baseline in Physician's Global Assessment (PGA) Score at Week 24
Description: PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity. A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity.
Time Frame: Baseline, 24 Weeks
Population: Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: Scores on a 3-point scale
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 28 | 28
Scores on a 3-point scale | -0.4 (0.09) | -0.4 (0.09)

18. Secondary Outcome: Mean Percent Change From Baseline in PGA Score at Week 24.
Description: The PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity. A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity.
Time Frame: Baseline, 24 weeks
Population: LOCF
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 28 | 28
Percentage | -26.1 (6.6) | -24.8 (13.1)

19. Secondary Outcome: Absolute Change From Baseline in the Safety of Estrogen in Lupus Erythematosus National Assessment SLE Disease Activity Index (SELENA SLEDAI) Score at Week 24
Description: SELENA SLEDAI is calculated from 24 individual descriptors; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare.
Time Frame: Baseline, 24 Weeks
Population: LOCF
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 28 | 28
Points on a scale | -2.9 (0.8) | -3.1 (0.5)

20. Secondary Outcome: Mean Percent Change From Baseline in the SELENA SLEDAI Score at Week 24
Time Frame: Baseline, 24 weeks
Population: LOCF
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 28 | 28
Percentage | -35.8 (9.1) | -40.5 (8.6)

21. Secondary Outcome: Absolute Change From Baseline in Complement C3 at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes only patients with low C3 (<900 mg/L) at baseline and must have had a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 5 | 10
mg/L | 188.0 (51.5) | 4.0 (44.3)

22. Secondary Outcome: Median Percent Change From Baseline in Compliment C3 at Week 24
Time Frame: Baseline, 24 Weeks
Population: as for outcome 21
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 5 | 10
Percentage | 25.8 [13.6 to 55.4] | 3.6 [-25.7 to 33.3]

23. Secondary Outcome: Absolute Change From Baseline in Complement C4 at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes only patients with low C4 (<16 mg/dL) at baseline and must have had a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 6 | 11
mg/dL | 7.2 (1.7) | 2.3 (1.4)

24. Secondary Outcome: Median Percent Change From Baseline in Complement C4 at Week 24
Time Frame: Baseline, 24 Weeks
Population: as for outcome 23
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 6 | 11
Percentage | 76.9 [0 to 133.3] | 40.0 [-46.7 to 200.0]

25. Secondary Outcome: Absolute Change From Baseline in Anti-Double-Stranded DNA (Anti-dsDNA)at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes only patients positive for anti-dsDNA (≥30 IU/mL) at baseline and must have had a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 11 | 14
IU/mL | -33.1 (11.1) | -6.0 (12.2)

26. Secondary Outcome: Median Percent Change From Baseline in Anti-dsDNA at Week 24
Time Frame: Baseline, 24 weeks
Population: as for outcome 25
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 11 | 14
Percentage | -24.0 [-51.4 to 18.4] | 0.0 [-57.2 to 125.8]

27. Secondary Outcome: Absolute Change From Baseline in High Density Lipoproteins (HDL) at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
mmol/L | 0.1 (0.04) | 0.0 (0.08)

28. Secondary Outcome: Median Percent Change From Baseline in HDL at Week 24
Time Frame: Baseline, 24 week
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
Percentage | 4.8 [-16.1 to 34.6] | 2.2 [-38.2 to 72.7]

29. Secondary Outcome: Absolute Change From Baseline in Total Cholesterol at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
mmol/L | 0.1 (0.09) | 0.0 (0.20)

30. Secondary Outcome: Median Percent Change From Baseline in Total Cholesterol at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
Percentage | 1.0 [-17.2 to 20.9] | 1.6 [-36.3 to 45.7]

31. Secondary Outcome: Median Percent Change From Baseline in Triglycerides at Week 24
Time Frame: Baseline, 24 weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Median (Full Range); unit: Percentage
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
Percentage | -4.9 [-46.9 to 183.0] | 4.5 [-59.4 to 120.6]

32. Secondary Outcome: Absolute Change From Baseline in Triglycerides at Week 24
Time Frame: Baseline, 24 Weeks
Population: Analysis population includes all patients with both a baseline and Week 24 laboratory sample.
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Number analyzed (Participants) | 25 | 24
mmol/L | -0.1 (0.14) | -0.0 (0.15)

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks
Groups:
- Belimumab SC Q2WKS: The Q2wk group will receive 100 mg of belimumab (1 injection) plus standard therapy on Days 0, 7, 14, and then every 2 weeks thereafter.
- Belimumab SC 3X/WK: The 3x/wk group will receive 200 mg of belimumab (2 injections of 100 mg each) plus standard therapy on Days 0, 2, and 4 and then 100 mg (1 injection) 3 times per week thereafter.
Arm/Group | Belimumab SC Q2WKS | Belimumab SC 3X/WK
Serious Adverse Events (participants affected / at risk) | 2/28 | 4/28
Other Adverse Events (participants affected / at risk) | 19/28 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab SC Q2WKS (N=28) | Belimumab SC 3X/WK (N=28)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belimumab SC Q2WKS (N=28) | Belimumab SC 3X/WK (N=28)
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 3 | 2
Injection site irritation (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 5 | 0
Sinusitis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
SLE arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center trials,no investigator will be authorized to publish study results from an individual center until the earlier of the multi-center trial results are published or 12 months after the end or termination of the multi-center trial at all sites. All manuscripts and abstracts must be submitted to the sponsor for review least 30 days prior to submission for publication or for presentation at a scientific meeting. The sponsor may delay publication for up to 3 months if indicated.